CLINICAL TRIAL: NCT02617277
Title: A Phase I Study Assessing the Safety, Tolerability and Pharmacokinetics of AZD1775 (Adavosertib) in Combination With MEDI4736 (Durvalumab) in Patients With Advanced Solid Tumours
Brief Title: Safety, Tolerability and Pharmacokinetics of AZD1775 (Adavosertib) Plus MEDI4736 (Durvalumab) in Patients With Advanced Solid Tumours
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6015C00002; REFMAL 412 (Other: Sarah Cannon Development Innovations, LLC)
Record Dates: First submitted 2015-11-26; First posted 2015-11-30 (Estimated); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumours
Keywords: AZD1775; MEDI4736; AZD1775 + MEDI4736; Advanced Solid Tumours; Adavosertib; Durvalumab
MeSH Terms: interventions — adavosertib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Schedule A (Experimental): In Schedule A, patients will receive MEDI4736 (durvalumab) by intravenous on Day 1, and AZD1775 (adavosertib) twice daily orally on Days 1-5 and Days 15-19 of a 28-day cycle. In all dose schedules, dexamethasone will be administered as an anti-emetic on the first day of the AZD1775 (adavosertib).
  Interventions: Drug: AZD1775; Drug: MEDI4736
- Dose Schedule B (Experimental): In Schedule B, patients will receive MEDI4736 (durvalumab) by intravenous on Day 1, and AZD1775 (adavosertib) twice daily orally on Days 15-17 and Days 22-24 of a 28-day cycle. In Schedule B there will be a 7-day AZD1775 (adavosertib) lead-in to enable serial PK measurements prior to initiating MEDI4736 on Day 1. In all dose schedules, dexamethasone will be administered as an anti-emetic on the first day of the AZD1775 (adavosertib) consecutive dosing day blocks including the lead-in portion of Schedules B, C, and D. Additional alternative dose levels and/or schedules may also be explored if emerging data suggest these would be more appropriate.
  Interventions: Drug: AZD1775; Drug: MEDI4736
- Dose Schedule C (Experimental): In Schedule C, patients will receive MEDI4736 (durvalumab) by intravenous on Day 1, and AZD1775 (adavosertib) twice daily orally on Days 8-10, Days 15-17, and Days 22-24 of a 28-day cycle. In Schedule C there will be a 7-day AZD1775 (adavosertib) lead-in to enable serial PK measurements prior to initiating MEDI4736 (durvalumab) on Day 1. In all dose schedules, dexamethasone will be administered as an anti-emetic on the first day of the AZD1775 (adavosertib) consecutive dosing day blocks including the lead-in portion of Schedules B, C, and D. Additional alternative dose levels and/or schedules may also be explored if emerging data suggest these would be more appropriate.
  Interventions: Drug: AZD1775; Drug: MEDI4736
- Dose Schedule D (Experimental): In Schedule D, patients will receive MEDI4736 (durvalumab) by intravenous on Day 1, and AZD1775 (adavosertib) one time per day orally on Days 15-19, and Days 22-26 of a 28-day cycle. In Schedule D there will be a 9-day lead-in period with AZD1775 (adavosertib) being dosed on Days -9 to -5 to enable serial PK measurements prior to initiating MEDI4736 (durvalumab) on Day 1. In all dose schedules, dexamethasone will be administered as an anti-emetic on the first day of the AZD1775 (adavosertib) consecutive dosing day blocks including the lead-in portion of Schedules B, C, and D. Additional alternative dose levels and/or schedules may also be explored if emerging data suggest these would be more appropriate.
  Interventions: Drug: AZD1775; Drug: MEDI4736

INTERVENTIONS:
Drug: AZD1775 — AZD1775 (adavosertib) is available in capsules for oral administration.
  Other Names: Adavosertib
Drug: MEDI4736 — MEDI4736 (durvalumab) will be administered by IV infusion.
  Other Names: Durvalumab

SUMMARY:
This study will assess the safety, tolerability, and pharmacokinetics of AZD1775 (adavosertib) given orally in combination with intravenous MEDI4736 (durvalumab). Secondly, the immunogenicity, pharmacodynamics, and preliminary anti-tumour activity will be determined in patients with refractory solid tumours.

DETAILED DESCRIPTION:
This is a Phase I, multi-center, dose-escalation study to assess the safety, tolerability and pharmacokinetics of oral therapy with AZD1775 (adavosertib) when combined with a fixed-dose of MEDI4736 (durvalumab). Immunogenicity, pharmacodynamics, and preliminary anti-tumour activity in patients with refractory solid tumours will also be investigated. In the initial design of this study a novel combination of AZD1775 (adavosertib) and MEDI4736 (durvalumab) was tested. The starting dose of AZD1775 (adavosertib) was 125 mg BID, over 5 days with 9 days off in 14-day cycles. This was designated Schedule A. This dose was not well tolerated. Two of six patients experienced dose limiting toxicity (DLT). The protocol was amended to include three additional dosing schedules. designated Schedules B, C, and D. In Schedule B patients will receive MEDI4736 (durvalumab) on Day 1, AZD1775 (adavosertib) on Days 15-17 and Days 22-24 of a 28-day cycle. In Schedule C, patients will receive MEDI4736 (durvalumab) on Day 1, AZD1775 (adavosertib) on Days 8-10, Days 15-17 and Days 22-24 of 28-day cycles. In Schedule D, patients will receive MEDI4736 (durvalumab) on Day 1 and AZD1775 (adavosertib) on Days 15-19 and Days 22-26 of a 28-day cycle. AZD1775 (adavosertib) will be dosed on a maximum of 6 days (Schedule B), 9 days (Schedule C), or 10 days (Schedule D) in each 28-day cycle. In all schedules, dexamethasone will be administered as an anti-emetic on the first day of each of the AZD1775 (adavosertib) consecutive dosing day blocks including the lead-in portion for Schedules B, C, and D. AZD1775 (adavosertib) will be administered at least 1 week after MEDI4736 (durvalumab) administration. Three to six patients will be enrolled in dose level 1 of Schedule B and evaluated for safety over a 28-day cycle prior to opening Schedule C dose level 1 for enrolment. Following safety evaluation of three to six patients in Schedule C dose level 1, a decision will be made by the Safety Review Team (SRT) to move forward with one or both schedules for further dose escalation. Three to six patients will be enrolled in Schedule D dose level 1 and evaluated for safety over a 28-day cycle. Patients in Schedule D will be evaluated for escalation independently of those in Schedules A, B, and C. Dose escalation will continue until identification of the Maximum Tolerated Dose (MTD). Once the MTD is determined this cohort will be expanded to a total of 18 patients to collect further safety data and for preliminary assessment of efficacy. Alternative dose levels/cohorts and/or schedules may be explored if emerging data suggest these would be more appropriate. The first day of Cycle 1 in Schedules B, C, and D will be preceded by a lead-in period of AZD1775 (adavosertib) monotherapy to enable serial sampling for assessment of pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving informed consent.
2. Males and females ≥18 years of age.
3. Weight ≥ 30 kg.
4. Histologic confirmation of a solid tumour, excluding lymphoma, refractory to standard therapy or for which no standard of care regimen exists.
5. Measurable or non-measureable disease according to RECIST v1.1.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
7. Baseline laboratory values within 7 days prior to receiving study drugs (without transfusion support):

   * Absolute neutrophil count (ANC) ≥1500/μL
   * Haemoglobin (HgB) ≥9 g/dL
   * Platelets ≥100,000/μL
   * Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2.5 x Upper Limit of Normal (ULN).
   * Serum bilirubin within normal limits (WNL) or ≤ 1.5 x ULN in patients with liver metastases; or total bilirubin ≤ 3.0 x ULN with direct bilirubin WNL in patients with well documented Gilbert's Syndrome.
   * Serum creatinine ≤ 1.5 x ULN, or creatinine clearance (CrCl) ≥ 40 mL/min as calculated by Cockcroft-Gault method.
8. Fertile females of child-bearing potential who agree to use adequate contraceptive measures from 2 weeks prior to the study and until 1 month after the last dose of AZD1775 (adavosertib) or 3 months after the last dose of MEDI4736 (durvalumab), whichever is later, who are not breastfeeding, and who have a negative serum or urine pregnancy test within 3 days prior to the start of study treatment.
9. Male patients must agree to use at least one medically acceptable form of contraception for the duration of the study and for 3 months after the last dose of AZD1775 (adavosertib) and MEDI4736 (durvalumab), whichever is later.
10. Predicted life expectancy ≥ 12 weeks.
11. Willing to provide consent for the collection of biological samples including circulating tumour DNA (ctDNA), and blocks or slides from archival diagnostic samples, or fresh tumour biopsy (if archival is not available) for analyses.
12. Willingness and ability to comply with study and follow-up procedures.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
2. Previous enrolment in this study.
3. Concurrent enrolment in another interventional clinical study.
4. Participation in another interventional clinical study or study with an investigational product during the last 28 days or 5 half-lives whichever is shorter.
5. Major surgical procedures (as defined by the Investigator) ≤28 days of beginning study treatment, or minor surgical procedures (as defined by the Investigator) ≤7 days. No waiting period required following Port-a-Cath placement. Note: Local surgery of isolated lesions for palliative intent is acceptable.
6. Palliative radiation therapy completed ≤ 7 days prior to start of study drugs.
7. No other anti-cancer therapy (chemotherapy, immunotherapy, hormonal anti-cancer radiotherapy [except for palliative local radiotherapy]), biological therapy or other novel agent is permitted while the patient is receiving study medication. Patients on luteinizing hormone-releasing hormone (LHRH) analogue treatment for more than 6 months are allowed entry into the study and can continue this treatment during the study.
8. Any unresolved NCI CTCAE Grade >1 toxicity from prior therapy (except alopecia or anorexia). Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with AZD1775 (adavosertib) or MEDI4736 (durvalumab) may be included after consultation with the Medical Monitor.
9. Inability to swallow oral medication.
10. Brain metastases or spinal cord compression unless the patient is stable (asymptomatic, no evidence of new or emerging brain metastases) and off steroids for at least 14 days prior to start of study treatment. Following radiotherapy and/or surgery, patients with brain metastases must wait 4 weeks following the intervention and must confirm stability with imaging before enrolment. Patients with suspected brain metastases at screening should have a CT/MRI of the brain prior to study entry. Brain metastases will not be recorded as RECIST target lesions (TL) at baseline.
11. History of leptomeningeal carcinomatosis.
12. Ascites requiring intervention (e.g. need for paracentesis or Tenckhoff catheter).
13. History of primary immunodeficiency.
14. History of tuberculosis.
15. Organ transplant that requires the use of immunosuppressive treatment.
16. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g. colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematous; sarcoidosis syndrome, or Wegner syndrome; Grave's disease; rheumatoid arthritis, hypophysitis, uveitis, etc.). The following are exceptions to this criterion: vitiligo or alopecia, hypothyroidism stable on hormone replacement, chronic skin condition that does not require treatment, patients without active disease in the last 5 years may be included after consultation with Medical Monitor, patients with celiac disease controlled by diet alone.
17. Any of the following cardiac diseases currently or within the last 6 months: unstable angina pectoris, congestive heart failure, acute myocardial infarction, heart failure ≥ 2 defined by NYHA, conduction abnormality not controlled with pacemaker or medication, significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible), history of Torsades de pointes unless all risk factors that contributed to Torsades have been corrected.
18. Uncontrolled hypertension.
19. Interstitial lung disease.
20. Known active cancers.
21. Mean resting corrected QT interval (specifically QTc calculated using the Fridericia formula [QTcF]) > 450 msec for males and > 470 msec for females from 3 ECGs performed within 2-5 minutes apart at study entry or congenital long QT syndrome.
22. Known serious active infection at study entry.
23. Serious chronic gastrointestinal conditions associated with diarrhoea within the past 12 months.
24. Pregnant or lactating.
25. Previous allogeneic bone marrow transplant.
26. Psychiatric illness or social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
27. Use of approved treatment (e.g. chemotherapy, targeted therapy, biologic therapy, or monoclonal antibody [mAb]) ≤ 21 days prior to the first dose of study drug. If there are questions relating to this criterion, a longer wash-out period may be required after discussion with the Medical Monitor.
28. Current or prior use of WEE-1 inhibitor or any immunosuppressive medication (e.g. anti-PDL1, anti-PD1, or previous cell-depleting therapies such as alemtuzumab, anti-CD4, anti-CD5, anti-CD3, anti-CD20, etc.) ≤ 14 days prior to the first dose of MEDI4736. The following are exceptions to this criterion: Intranasal, inhaled, topical, or local steroid injections (e.g. intra-articular injection), systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent. Please note: This does not include use of corticosteroids as part of antiemetic prophylaxis or treatment in relation to AZD1775 (adavosertib) dosing or steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication).
29. Any known allergy, hypersensitivity or contraindication to the components of the study drug AZD1775 (adavosertib) or MEDI4736 (durvalumab) or any of their excipients, or to corticosteroids.
30. Prior randomisation in a previous MEDI4736 (durvalumab) clinical study regardless of treatment arm assignment.
31. Receipt of live attenuated vaccine ≤ 30 days prior to the first dose of study drug. Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
32. Prescription or non-prescription drugs or other products known to be sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors or inducers of CYP3A4 which cannot be discontinued 2 weeks prior to the first day of study drug dosing and withheld throughout the study until 2 weeks after the last dose of study drug.
33. Herbal preparations must be stopped 7 days prior to first dose of study drug.
34. Any evidence of severe or uncontrolled systemic disease such as active bleeding diatheses (as judged by the Investigator), or positive for immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV).
35. Non-leukocyte depleted whole blood transfusion within 120 days of genetic sample collection.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-12-28 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of Dose Limiting Toxicities (DLTs) | Up to 28 Days
  DLTs are defined as:
  1. Grade 4 haematologic toxicity for ≥7 days, including infection with febrile neutropenia, or Grade 4 thrombocytopenia.
  2. Grade 3 thrombocytopenia associated with Grade ≥2 bleeding.
  3. Non-haematologic toxicity ≥Grade 3.
  4. Grade 3 nausea, vomiting, or diarrhoea that does not respond within 48 hours.
  5. Grade 4 nausea, vomiting, and diarrhoea.
  6. ALT or AST ≥5 x but ≤8 x ULN that does not resolve to Grade 2 within 5 days. ALT or AST >8 x ULN or total bilirubin >5 x ULN is a DLT regardless of duration.
  7. AST or ALT >3 x ULN and concurrent increase in total bilirubin > 2 x ULN (Hy's Law) without evidence of cholestasis or alternative explanations (viral hepatitis, disease progression in the liver).
  8. Grade ≥2 pneumonitis that does not resolve to ≤ Grade 1 within 7 days.
  9. Clinically significant or unacceptable toxicity that does not respond to supportive care, or results in a disruption of dosing for >7 days.

SECONDARY OUTCOMES:
The incidence and severity of treatment emergent adverse events (TEAEs) graded according to NCI CTCAE v4.03 | Throughout the study (approximately 18 months).
Change from baseline in physical examination findings | Throughout the study (approximately 18 months).
  A complete physical examination will be performed on Day 1 of each cycle and at the End-of-Treatment (EOT) visit. The examination will include an assessment of general appearance; abdomen, skin, head and neck; lymph nodes, and thyroid; and respiratory, cardiovascular, musculoskeletal and neurological systems.
Change from baseline in clinical chemistry, hematology, and coagulation parameters | Throughout the study (approximately 18 months).
  Blood samples for monitoring of clinical chemistry parameters and determination of haematology will be taken at screening, Days 1, 8, 15, and 22 of Cycle 1, Days 1, 8, and 15 of each cycle thereafter, and at the end-of-treatment visit.
Change from baseline in vital signs | Throughout the study (approximately 18 months).
  Resting heart rate, blood pressure, respiration rate, temperature, and weight at the screening visit. Height will be measured at the screening visit only. Vital signs and weight should be obtained Day 1 of each treatment cycle and at the EOT visit.
Determine the presence of Anti-Drug Antibodies (ADA) to MEDI4736 (durvalumab). | Throughout the study (approximately 18 months).
  The presence of Anti-Drug Antibodies (ADA) to MEDI4736 (durvalumab) will be determined as a measure of the immunogenicity of MEDI4736 in combination with AZD1775 (adavosertib).
Objective Response Rate (ORR) | Estimated 18 months
  The preliminary anti-tumour activity of AZD1775 (adavosertib) when combined with MEDI4736 (durvalumab) in patients with advanced solid tumours will be determined by the Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
  The objective response rate (ORR) is defined as the number of the patients with a confirmed best overall response of Complete Response (CR) or Partial Response (PR) divided by the number of patients in the efficacy analysis set.
Progression-Free Survival (PFS) | Estimated 18 months
  The preliminary anti-tumour activity of AZD1775 (adavosertib) when combined with MEDI4736 (durvalumab) in patients with advanced solid tumours will be determined by the Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
  Progression-free survival (PFS) is defined as the time from date of first dose of MEDI4736 until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from therapy or receives another anti-cancer therapy prior to progression. Patients who have not progressed or died at the time of analysis will be censored at the latest date of assessment from their last evaluable RECIST assessment.
Disease Control Rate (DCR) | Estimated 18 months
  The preliminary anti-tumour activity of AZD1775 (adavosertib) when combined with MEDI4736 (durvalumab) in patients with advanced solid tumours will be determined by the Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
  The disease control rate (DCR) is defined as the percentage of patients in the efficacy analysis set with a confirmed best overall response of CR or PR, or a best overall response of Stable Disease (SD).
Overall Survival (OS) | Estimated 18 months
  The preliminary anti-tumour activity of AZD1775 (adavosertib) when combined with MEDI4736 (durvalumab) in patients with advanced solid tumours will be determined by the Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
  Overall survival is defined as the time from the date of first dose of study drug until death due to any cause. Any subject known to be alive at the time of analysis will be censored based on the last recorded date on which the subject was known to be alive. Equivalent to PFS, patients will be followed for survival until the last patient has discontinued study drug.
QTc interval | Up to 28 days
  To characterise the effect of AZD1775 (adavosertib) on QTc in patients with advanced solid tumours when combined with MEDI4736 (durvalumab) triplicate ECGs will be obtained at screening and approximately 2-5 minutes apart at the time of PK sample collection as follows: Day -5 pre-dose AZD1775 (adavosertib), Cycle 1 Day 17 pre-dose AZD1775 (adavosertib) and 4 hours post-dose. The ECG assessments will be performed before the PK sample is collected.
Levels of immunologically relevant leukocyte subpopulations | Up to 28 days
  Levels of immunologically relevant leukocyte subpopulations will be measured by analysis of a panel of cytokines and chemokines involved in Th1-driven immune responses and changes in proliferating T cells.
Plasma concentrations of AZD1775 (adavosertib) and MEDI4736 (durvalumab) when given in combination, and of AZD1775 (adavosertib) when given alone. | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Manish Patel, M.D., Principal Investigator — Florida Cancer Specialists
Locations (3):
- United States (3):
  - Research Site, Denver, Colorado
  - Research Site, Sarasota, Florida
  - Research Site, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Patel MR, Falchook GS, Wang JS, Imedio ER, Kumar S, Miah K, Mugundu GM, Jones SF, Spigel DR, Hamilton EP. Open-Label, Multicenter, Phase I Study to Assess Safety and Tolerability of Adavosertib Plus Durvalumab in Patients with Advanced Solid Tumors. Target Oncol. 2025 Jan;20(1):127-138. doi: 10.1007/s11523-024-01110-8. Epub 2024 Nov 19. PMID 39560862